CLINICAL TRIAL: NCT04368286
Title: Effects of Respiratory Rehabilitation on Patients After Extubation
Brief Title: Effects of Respiratory Rehabilitation on ICU Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2018-212-01
Record Dates: First submitted 2020-04-22; First posted 2020-04-29 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: ICU Acquired Weakness; Rehabilitation
Keywords: ICU，rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation group (Experimental): To conduct a comprehensive pulmonary rehabilitation assessment and treatment
  Interventions: Behavioral: pulmonary rehabilitation
- Conventional medical group (No Intervention): Conventional medical treatment

INTERVENTIONS:
Behavioral: pulmonary rehabilitation — Pulmonary rehabilitation (respiratory rehabilitation) is a comprehensive intervention based on a comprehensive patient assessment, targeted to the treatment of patients, including but not limited to exercise training, education and behavior change, aimed at improving the physical and mental health of patients with chronic respiratory diseases and promoting long-term adherence to health-enhancing behaviors.
  Arms: Rehabilitation group

SUMMARY:
Effects of respiratory rehabilitation on patients after extubation

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether sequential treatment with high-flow humidification therapy apparatus can improve the postoperative recovery and functional status of patients with invasive mechanical ventilation in ICU after the withdrawal of the catheter.Inclusion criteria: age 18-95;The hemodynamics were stable, that is, 50 < heart rate less than 120 beats/min, 90 < systolic blood pressure < 200mmHg, 55 < mean arterial pressure < 120mmHg.Do not increase the dose of vasopressor for at least 2 hours;Intracranial pressure was stable and there was no seizure within 24 hours.The breathing condition was stable, that is, the oxygen satiety of the patient's finger vein was ≥88%, and the breathing frequency was >10 and< 35 times/min.Exclusion criteria: pregnancy;Acute myocardial infarction.A total of 50 patients who are sequentially treated with high-flow humidification therapy apparatus after extubation in ICU are randomly assigned. The experimental group receive respiratory rehabilitation therapy, while the control group only receive routine medical treatment. All the enrolled patients underwent rehabilitation evaluation and bedside diaphragmatic ultrasound measurement.This study was approved by the Ethics Committee of the CPLA General Hospital (project No.2018-212-01). The following clinical datas were recorded for all patients through the unified database software: The rehabilitation program was formulated according to the cluster management strategy of ABCDEF and the six-step method of early activities.All of the patients in monitoring vital signs, every day at hospital group and all peripheral muscle MRC assessment, 30 s sit stand trial, modified Barthel index, Borg dyspnea score, arterial blood gas analysis, diaphragm ultrasonic monitoring by the bed, finally the experimental process on the patients whether using noninvasive ventilator, whether for endotracheal intubation again, whether to have new complications (pressure sores, aspiration, thrombosis, etc.) and the patients bed time statistics for the first time. Statistical analyses were conducted by SPSS 21.0 and a two-tailed P < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18
* The hemodynamics are stable
* 50 < heart rate less than 120 beats/min
* 90 < systolic blood pressure < 200mmHg
* 55 < mean arterial pressure < 120mmHg
* Do not increase the dose of vasopressor for at least 2 hours
* Intracranial pressure was stable and there is no seizure within 24 hours
* The breathing condition is stable
* the oxygen satiety of the patient's finger vein is ≥88%
* 10<the breathing frequency < 35 times/min

Exclusion Criteria:

* Pregnancy
* Acute myocardial infarction (ami)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-20 (Estimated); Primary Completion 2021-04-20 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
Reintubation rates | 28 days
  The artificial airway was established again for invasive mechanical ventilation

SECONDARY OUTCOMES:
MRC，medical research council | 28 days
  medical research council，Assessment of peripheral muscle strength，total points0~60，less than 48scores means ICU aquired weaknesses.
30-STS | 28 days
  30 second sit-to-stand test.The more times, has the better muscular endurance.
Barthel | 28 days
  Assessment of activities of daily living.total points0~100，less than 60 scores means can't independent living.
Borg dyspnea score | 28 days
  total points0~10,The higher the grade, the more difficulty breathing.
oxygen partial pressure | 28 days
  Partial pressure of oxygen in arterial blood,normal range is 80~100.
oxygenation index | 28 days
  The partial pressure of oxygen divided by the concentration of oxygen,Normal is greater than 400.
The diaphragmatic excursion | 28 days
  The distance the diaphragm moves up and down during breathing,normal is 1.4cm.
diaphragm contraction rate | 28 days
  The rate at which the diaphragm contracts during breathing,normal is 1.3cm/s.
diaphragm thickness diaphragm thickness fraction | 28 days
  Thickness of diaphragm during breathing,(Diaphragm thickness at the end of inhalation-Diaphragm thickness at the end of exhalation)/Diaphragm thickness at the end of exhalation
length of stay in ICU | three months
  Length of stay in ICU
LOS(length of stay) | three months
  length of stay in hospital
First time out of bed | three months
  First time out of bed by oneself
Noninvasive utilization rate | 28 days
  Non-invasive ventilator usage
mortality | 28 days
  Alive or Dead
Complication rate | 28 days
  The incidence of new complications(pressure sores、thrombus、aspiration)

CONTACTS AND LOCATIONS:
Overall Officials: xin li xie, Ph.D., Principal Investigator — Study Principal Investigator Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464